CLINICAL TRIAL: NCT00163020
Title: 17-Alpha-Hydroxyprogesterone Caproate for Reduction of Neonatal Morbidity Due to Preterm Birth in Twin and Triplet Pregnancies - A Concurrent Randomized Double-blinded Clinical Trial
Brief Title: 17OHP for Reduction of Neonatal Morbidity Due to Preterm Birth (PTB) in Twin and Triplet Pregnancies
Acronym: 170HP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Obstetrix Medical Group (Industry)
Responsible Party: Sponsor
Organization: Pediatrix (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OBX0003; OBX 0012 (Other: Obstetrix CREQ Protocol Number)
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Results first posted 2012-11-07 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Preterm Birth
Keywords: Preterm Birth; Preterm Delivery; Multiple gestation; 17-alpha-hydroxyprogesterone caproate; Progesterone
MeSH Terms: conditions — Premature Birth | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Test Group (170HP) (Active Comparator): Test Group will receive weekly doses of 170HP via injection as early as 19weeks until 34.0weeks gestation or delivery which ever comes first.
  Interventions: Drug: 17-alpha-hydroxyprogesterone caproate injectable
- 2 - Control (Normal Saline) (Placebo Comparator): Control Group will receive weekly doses of placebo (NS) via injection as early as 19weeks until 34.0weeks gestation or delivery which ever comes first.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 17-alpha-hydroxyprogesterone caproate injectable — 250mg of 17-alpha-hydroxyprogesterone caproate (+ preservatives) injectable weekly starting as early as 19wks gestation until 34.0wks gestation of delivery which ever comes first.
  Other Names: 170HP
  Arms: 1 Test Group (170HP)
Drug: Placebo — Weekly doses of placebo (NS + preservatives) via injection as early as 19weeks until 34.0weeks gestation or delivery which ever comes first.
  Other Names: Normal Saline
  Arms: 2 - Control (Normal Saline)

SUMMARY:
Hypothesis: Among women with twin or triplet pregnancies, weekly injections of 17-alpha-hydroxyprogesterone caproate (17OHP), started before 24 weeks of gestation, will reduce neonatal morbidity by reducing the rate of preterm delivery.

This study involves two concurrent double-blinded randomized clinical trials of 17OHP versus placebo. Each trial will test the efficacy and safety of 17OHP in women with a specific risk factor for preterm birth. The two risk factors to be studied are:

1. Twin pregnancy
2. Triplet pregnancy

DETAILED DESCRIPTION:
Prematurity is a leading cause of neonatal morbidity and mortality in the USA. Nationally, 12% of all babies deliver before term and 3% deliver before 32 wks gestational age (GA). Recent studies suggest that 17OHP and other progesterone derivatives may reduce the rate of preterm birth among women with a history of prior preterm birth. However, it has not been demonstrated that this reduction in preterm birth is accompanied by a clinically significant reduction in neonatal complications. Further, most women who deliver preterm have no history of a prior preterm birth. Little is known about whether progesterone treatment is effective in women with other risk factors for preterm birth such as multiple gestation. The proposed study will assess the role of 17OHP in women with twin or triplet pregnancies and will assess the impact on neonatal health, not merely the impact on gestational age at delivery. Prior studies were not designed to be large enough to have statistical power to assess effects on neonatal morbidity.

In the 6 trials combined in the Goldstein meta-analysis, only 279 women were treated with 17OHP and only 73 women had a preterm delivery. The NICHD study presented by Meis approximately doubles the world-wide experience, with 306 women under treatment, of whom 73 delivered prior to 35 wks. Yet, this study was not designed to have power to show a reduction in neonatal complications but only a reduction in preterm birth rates.

The present study is the first to be specifically designed to have adequate power to test whether 17OHP reduces neonatal morbidity among women with one of two specific risk factors for preterm birth.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age (GA) 15-23w0d gestational age at the time of recruitment
2. GA 16w0dk to 23w6d at the time of randomization and initiation of injections
3. Maternal age 18 years or older
4. One of these risk factors for spontaneous preterm birth:

   1. Twins in current pregnancy, dichorionic placentation
   2. Triplets in current pregnancy, trichorionic placentation
5. Intact membranes
6. Patient has had at least one detailed 2nd-trimester ultrasound examination documenting placentation, chorionicity, fetal number, fetal size, amniotic fluid volumes, and fetal anatomy. (This examination must comply with minimum standards such as those published by the American Institute of Ultrasound in Medicine, American College of Radiology, or American College of Obstetricians & Gynecologists It is NOT mandatory that this examination be performed at the research-study center.)
7. Investigator believes patient will be reliable with follow-up visits and believes that delivery data and neonatal data are likely to be available.

Exclusion Criteria:

1. Symptomatic uterine contractions in current pregnancy
2. Contraindication to interventions intended to prolong the pregnancy (including lethal fetal anomalies, amnionitis, preeclampsia, severe oligohydramnios, severe growth delay, fetal death appears imminent or inevitable)
3. Risk factors for major neonatal morbidity unrelated to preterm delivery (such as monochorionic placentation in multiple gestation, major malformations, certain medication exposures)
4. Preexisting maternal medical condition that might be worsened by progesterone therapy, including: asthma requiring medications, renal insufficiency, seizure disorder, ischemic heart disease, active cholecystitis, impaired liver function, history of thromboembolic disorder, history of breast cancer, history of major depression requiring hospitalization.
5. Preexisting maternal medical condition associated with a high risk of preterm delivery including: refractory hypertension, diabetes with nephropathy or retinopathy, renal insufficiency, active systemic lupus erythematosus. Note that a history of prior preterm birth is NOT an exclusion.
6. Use of progesterone or progesterone-derivative medication after 15 weeks gestation in current pregnancy.
7. Allergy to 17OHP or oil vehicle.
8. Placement of emergent cerclage (defined as one placed after the occurrence of cervical change such as dilation, funneling, or effacement) with this pregnancy. Prophylactic cerclage is NOT an exclusion (defined as one placed before any cervical change, for example, because of a history of cervical incompetence, or because of a prior cervical procedure such as LEEP or cone biopsy).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2004-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Maurel, RN, MSN, CNS, Study Director — Obstetrix Medical Group, Inc.; Andrew Combs, MD, Principal Investigator — Obstetrix Medical Group, Inc.
Locations (18):
- United States (18):
  - Banner Good Samaritan Hospital, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Saddleback Memorial Medical Center, Laguna Hills, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - University of Southern California-Irvine Medical Center, Orange, California
  - Good Samaritan Hospital, San Jose, California
  - Swedish Medical Center, Denver, Colorado
  - Presbyterian/St Luke's Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Skyridge Medical Center, Lonetree, Colorado
  - Mercy Medical Center, Des Moines, Iowa
  - Saint Luke's Hospital, Kansas City, Kansas City, Missouri
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Harris Methodist Fort Worth Hospital, Fort Worth, Texas
  - Evergreen Hospital, Kirkland, Washington
  - Swedish Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goldstein P, Berrier J, Rosen S, Sacks HS, Chalmers TC. A meta-analysis of randomized control trials of progestational agents in pregnancy. Br J Obstet Gynaecol. 1989 Mar;96(3):265-74. doi: 10.1111/j.1471-0528.1989.tb02385.x. PMID 2653414
- [Background] da Fonseca EB, Bittar RE, Carvalho MH, Zugaib M. Prophylactic administration of progesterone by vaginal suppository to reduce the incidence of spontaneous preterm birth in women at increased risk: a randomized placebo-controlled double-blind study. Am J Obstet Gynecol. 2003 Feb;188(2):419-24. doi: 10.1067/mob.2003.41. PMID 12592250
- [Background] Meis PJ, Klebanoff M, Thom E, Dombrowski MP, Sibai B, Moawad AH, Spong CY, Hauth JC, Miodovnik M, Varner MW, Leveno KJ, Caritis SN, Iams JD, Wapner RJ, Conway D, O'Sullivan MJ, Carpenter M, Mercer B, Ramin SM, Thorp JM, Peaceman AM, Gabbe S; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Prevention of recurrent preterm delivery by 17 alpha-hydroxyprogesterone caproate. N Engl J Med. 2003 Jun 12;348(24):2379-85. doi: 10.1056/NEJMoa035140. PMID 12802023
- [Background] American College of Obstetricians & Gynecologists. Special problems of multiple gestation. Educational Bulletin 253, 1998.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential women carrying a twin or triplet pregnancy meeting defined inclusion and exclusion criteria were recruited from participating outpatient medical clinics from November, 2004 to August 2009.
Pre-assignment Details: During the pre-assignment period, subjects were consented to participate, giving a compliance injection of Castor Oil and brought back 5 to 9 days later for re-evaluation. Exclusions were made based on the presence of a reaction to the injection, not meeting inclusion/exclusion criteria or the participates desire not to participate.
Groups:
- 1 Test Group (170HP): Test Group will receive a weekly dose of 170HP via injection as early as 19weeks until 34weeks 0days gestation or delivery which ever comes first.
- 2 - Control (Castor Oil): Control Group will receive a weekly dose of placebo (castor oil) via injection as early as 19weeks until 34weeks 0days gestation or delivery which ever comes first.
Period: Overall Study
Arm/Group | 1 Test Group (170HP) | 2 - Control (Castor Oil)
Started | 216 (Twins = 160 Triplets = 56) | 105 (Twins = 80 Triplets = 25)
Completed | 216 (Twins = 160 Triplets = 56) | 103 (Twins = 78 Triplets = 25)
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Test Group (170HP) | 2 - Control (Castor Oil) | Total
Number analyzed (Participants) | 216 | 105 | 321
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 216 | 105 | 321
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  twins | 34.0 (5.8) | 34.5 (6.6) | 34.3 (6.2)
  triplets | 33.4 (5.0) | 33.6 (5.4) | 33.5 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 105 | 321
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 216 | 105 | 321

OUTCOME MEASURES:

1. Primary Outcome: Newborn Respiratory Distress Syndrome (RDS)
Description: Newborn RDS in the twin arm is defined as compatible symptoms with radiographically confirmed hyaline membrane disease or with respiratory insufficiency of prematurity requiring ventilator support.
  Data expressed as mean n(%),Odds ratio, CI, and P-value were determined using repeated measures model wherein each twin/triplet within a given pregnancy is considered a repeated measure. Exceptions are comparison with 0 outcomes in one or both groups, so Fisher's Exact Test was used.
  Morbidity measures were based on live births with data available for the outcomes.
Time Frame: Measured from delivery until 30 days after baby was discharged from the hospital
Population: Population analysed were total Twin infants delivered to mothers within each study arm. (ie. babies born to moms in active arm (319) vs. babies born to mothers in placebo arm(153))
Measure: Number; unit: Twins
Groups:
- Twins Group = Test Arm - 17OHP: Weekly injection of 170HP (250mg)to patients with Twin Pregnancies
- Twins Group - Placebo Arm: Weekly injection of Placebo medication (castor oil)to patients with Twin Pregnancies
Arm/Group | Twins Group = Test Arm - 17OHP | Twins Group - Placebo Arm
Number analyzed (Participants) | 319 | 153
Twins | 44 [0.6 to 2.6] | 18 [0.6 to 2.6]

2. Primary Outcome: Use of Oxygen Therapy at 28 Days of Newborn Life
Description: Supplemental oxygen use by the baby measured at the point that the baby reaches 28 days old (after birth)within the twin group.
Time Frame: Measured at 28 days after birth.
Population: Population analysed were total Twin infants delivered to mothers within each study arm. (ie. babies born to moms in active arm (308) vs. babies born to mothers in placebo arm(150))
Measure: Number; unit: Twins
Arm/Group | Twins Group = Test Arm - 17OHP | Twins Group - Placebo Arm
Number analyzed (Participants) | 308 | 150
Twins | 9 | 0

3. Primary Outcome: Newborn Sepsis
Description: Newborn Sepsis in the twin group was defined as the presence of positive blood culture obtained in the first week of life in association with clinical findings suggesting illness for which the neonate received antibiotics.
Time Frame: measured during the first week following birth
Population: The participants were randomized in a two to one fashion (2=active participants to every 1=placebo participant). The number of participated included were based on an intent to treat protocol.
Measure: Number; unit: participants
Arm/Group | Twins Group = Test Arm - 17OHP | Twins Group - Placebo Arm
Number analyzed (Participants) | 319 | 154
participants | 3 | 1

4. Primary Outcome: Newborn Pneumonia
Description: Newborn Pneumonia in the twin group is described as compatible symptoms with diagnostic radiograph findings and positive results on blood cultures, persistent leukopenia
Time Frame: measure during the first 28 days after birth.
Population: Population analysed were total Twin infants delivered to mothers within each study arm. (ie. babies born to moms in active arm (320) vs. babies born to mothers in placebo arm(154))
Measure: Number; unit: Twins
Arm/Group | Twins Group = Test Arm - 17OHP | Twins Group - Placebo Arm
Number analyzed (Participants) | 320 | 154
Twins | 1 | 0

5. Primary Outcome: Newborn Intraventricular Hemorrhage Grade 3 or 4
Description: Newborn Intraventricular hemorrhage (IVH) Stage III in the twin group is described as - IVH with ventricular dilatation.
  Neonatal Intraventricular hemorrhage (IVH)Stage IV in the twin group is described as - IVH with parenchymal extension.
Time Frame: measured during the first 28 days after birth
Population: Population analysed were total Twin infants delivered to mothers within each study arm. (ie. babies born to moms in active arm (316) vs. babies born to mothers in placebo arm(152))
Measure: Number; unit: Twins
Arm/Group | Twins Group = Test Arm - 17OHP | Twins Group - Placebo Arm
Number analyzed (Participants) | 316 | 152
Twins | 3 | 0

6. Primary Outcome: Newborn Periventricular Leukomalacia (PVL)
Description: Newborn Periventricular leukomalacia (PVL) in the twin group is described as the presence of more than 1 obvious hypo echoic cyst in the periventricular white matter.
Time Frame: measured in the first 28 days after birth.
Population: The participants were randomized in a two to one fashion (2=active participants to every 1=placebo participant). The number of participants for analysis was determined using an intention to treat protocol.
Measure: Number; unit: participants
Arm/Group | Twins Group = Test Arm - 17OHP | Twins Group - Placebo Arm
Number analyzed (Participants) | 316 | 151
participants | 1 | 1

7. Primary Outcome: Newborn Necrotizing Enterocolitis (NEC)Requiring Surgery
Description: Newborn NEC in the twin group is described as the presence of any of the following: (1)unequivocal intramural air in abdominal radiograph; (2) perforation abdominal radiograph; (3) clinical evidence of perforation (erythema and induration of the abdominal wall or intrabdominal abscess formation); (4) characteristic findings observed at surgery or autopsy; (5) Stricture formation after an episode of suspected necrotizing enterocolitis.
Time Frame: measured in the first 28 days after birth
Population: Population analysed were total Twin infants delivered to mothers within each study arm. (ie. babies born to moms in active arm (315) vs. babies born to mothers in placebo arm(152))
Measure: Number; unit: Twins
Arm/Group | Twins Group = Test Arm - 17OHP | Twins Group - Placebo Arm
Number analyzed (Participants) | 315 | 152
Twins | 0 | 0

8. Primary Outcome: Newborn Retinopathy of Prematurity (ROP)
Description: Newborn ROP within the twin group is described as retinopathy confirmed on fundoscopic examination, felt to be due to prematurity and subsequent oxygen therapy.
Time Frame: measured during the first 28 day after birth
Population: Population analysed were total Twin infants delivered to mothers within each study arm. (ie. babies born to moms in active arm (308) vs. babies born to mothers in placebo arm(145))
Measure: Number; unit: Twins
Arm/Group | Twins Group = Test Arm - 17OHP | Twins Group - Placebo Arm
Number analyzed (Participants) | 308 | 145
Twins | 2 | 0

9. Primary Outcome: Newborn Asphyxia With Ischemic Injury of Brain, Heart, Kidneys, or Liver
Description: Newborn Asphyxia or Hypoxic-ischemic encephalopathy (HEI) within the twin group is characterized by clinical and laboratory evidence of acute or subacute brain injury due to asphyxia (ie, hypoxia, acidosis).
Time Frame: measured during the first 28 days after delivery
Population: Population analysed were total Twin infants delivered to mothers within each study arm. (ie. babies born to moms in active arm (274) vs. babies born to mothers in placebo arm(130))
Measure: Number; unit: Twins
Arm/Group | Twins Group = Test Arm - 17OHP | Twins Group - Placebo Arm
Number analyzed (Participants) | 274 | 130
Twins | 0 | 0

10. Secondary Outcome: Individual Components of Neonatal Morbidity (RDS, IVH-III/IV, Bronchopulmonary Dysplasia(BPD), PVL, Sepsis, NEC, ROP-Stage 3/4, Perinatal Death)
Description: Composite Neonatal Morbidity within the twin group is described as the presence of any one or more of the following neonatal morbidities (RDS, IVH-III/IV, BPD, PVL, sepsis, NEC, ROP-Stage 3/4, Perinatal Death).
Time Frame: measured as any event noted in the first 28 day following birth.
Population: Population analysed were total Twin infants delivered to mothers within each study arm. (ie. babies born to moms in active arm (320) vs. babies born to mothers in placebo arm(155))
Measure: Number; unit: Twins - Components of Neonatal Morbidity
Arm/Group | Twins Group = Test Arm - 17OHP | Twins Group - Placebo Arm
Number analyzed (Participants) | 320 | 155
Twins - Components of Neonatal Morbidity | 46 | 19

11. Secondary Outcome: Twins: Delivery Prior to 28 Weeks (Wks), 32 Wks, 34wks, and 37 Wks
Description: Gestational age was noted at time of delivery and stratified into three categories (Twins: Delivery prior to 28 weeks (wks), 32 wks, 34 wks, and 37 wks)
Time Frame: Gestational age noted at time of birth
Population: Population analysed were total pregnancies of mothers with twin gestation (ie. active group 160 and placebo group 80)
Measure: Number; unit: Twin Pregnancies
Arm/Group | Twins Group = Test Arm - 17OHP | Twins Group - Placebo Arm
Number analyzed (Participants) | 160 | 80
Twin Pregnancies
  Delivery before 28 weeks of gestation | 3 | 1
  Delivery before 32 weeks of gestation | 15 | 4
  Delivery before 34 weeks of gestation | 31 | 11
  Delivery before 37 weeks of gestation | 113 | 46

12. Secondary Outcome: Triplets: Delivery Prior to 28 Wks, 32 Wks, 35 Wks
Description: Gestational age was noted at time of delivery and stratified into three categories (Triplets: Delivery prior to 28 wks, 32 wks, 35 wks)
Time Frame: noted at delivery
Population: Population analysed were total pregnant mothers with triplet gestations (ie. active group 160 and placebo group 80)
Measure: Number; unit: Triplet Pregnancies
Groups:
- Triplet Group = Test Arm - 17OHP: Weekly injection of 170HP (250mg)to patients with Triplet Pregnancies
- Triplet Group - Placebo Arm: Weekly injection of Placebo medication (castor oil)to patients with Triplet Pregnancies
Arm/Group | Triplet Group = Test Arm - 17OHP | Triplet Group - Placebo Arm
Number analyzed (Participants) | 56 | 25
Triplet Pregnancies
  Delivery before 28 weeks of gestation | 9 | 2
  Delivery before 32 weeks of gestation | 19 | 13
  Delivery before 35 weeks of gestation | 43 | 13

13. Secondary Outcome: Newborn Gestational Age (GA) at Delivery
Description: Newborn Gestational age at delivery within the twin group is described as the gestational age of the baby on the day of birth.
Time Frame: determined at the time of birth
Population: Population analysed were total pregnant mothers with twin gestations (ie. active group 160 and placebo group 80)
Measure: Mean (Standard Deviation); unit: weeks of age for twin pregnancy
Arm/Group | Twins Group = Test Arm - 17OHP | Twins Group - Placebo Arm
Number analyzed (Participants) | 160 | 80
weeks of age for twin pregnancy | 35.3 (2.5) | 35.9 (2.3)

14. Secondary Outcome: Newborn Birthweight
Description: Newborn Birthweight within the twins group was measure following delivery and noted in grams.
Time Frame: measure following delivery
Population: Population analysed were twins from twin pregnancies (ie. active group 160 and placebo group 80)
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Twins Group = Test Arm - 17OHP | Twins Group - Placebo Arm
Number analyzed (Participants) | 160 | 78
grams | 2321 (523) | 2469 (543)

15. Secondary Outcome: Participant Drop-out Rates
Description: Drop-out rates in the twin group are described as any randomized participant who is withdrawn from the trial between randomization (as early at 16 weeks of pregnancy) and completion of the final dose of study medication (as late as 34 weeks of pregnancy).
Time Frame: any time from randomization to completion of final dose of study medication
Population: Population analysed were total pregnant mothers (participants) with twin gestation (ie. active group 160 and placebo group 80)
Measure: Number; unit: participants
Arm/Group | Twins Group = Test Arm - 17OHP | Twins Group - Placebo Arm
Number analyzed (Participants) | 160 | 80
participants | 8 | 5

16. Secondary Outcome: Participant Side Effects Requiring Cessation of Therapy
Description: Describe as the cessation of study related therapy for the participant within the twin group at anytime from initial study related injection until the final injection at 34 weeks of pregnancy.
Time Frame: anytime from initial injection to final injection at 34 weeks.
Population: as for outcome 15
Measure: Number; unit: participants
Arm/Group | Twins Group = Test Arm - 17OHP | Twins Group - Placebo Arm
Number analyzed (Participants) | 160 | 80
participants | 6 | 0

17. Primary Outcome: Perinatal Death
Description: Perinatal death within the twin group is described as a stillbirth, neonatal death, or miscarriage after randomization.
Time Frame: measured from randomization to 28 days after birth.
Population: Population analysed were total Twin infants delivered to mothers within each study arm. (ie. babies born to moms in active arm (320) vs. babies born to mothers in placebo arm(156))
Measure: Number; unit: Twins
Arm/Group | Twins Group = Test Arm - 17OHP | Twins Group - Placebo Arm
Number analyzed (Participants) | 320 | 156
Twins | 0 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 4.9 years the trial was actively enrolling subjects. For each randomized participant, adverse events were captured from randomization until the participant and her baby were discharged from the hospital.
Description: Assessments were both Systematic & Non-systematic: standard questionnaire, regular investigator assessment, regular laboratory testing, systematic evaluation of medical record, self-reporting by participants, occasional assessment/testing
Groups:
- Test Group (170HP): Both Twins and Triplets in the Test Group received a weekly dose of 170HP via injection as early as 19weeks until 34weeks 0days gestation or delivery which ever came first.
- Control (Castor Oil): Both Twins and Triplets in the Control Group received a weekly dose of placebo (castor oil) via injection as early as 19weeks until 34weeks 0days gestation or delivery which ever came first.
Arm/Group | Test Group (170HP) | Control (Castor Oil)
Serious Adverse Events (participants affected / at risk) | 69/216 | 34/105
Other Adverse Events (participants affected / at risk) | 40/216 | 18/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Group (170HP) (N=216) | Control (Castor Oil) (N=105)
Postpartum Hemorrhage requiring blood transfusion (Pregnancy, puerperium and perinatal conditions) | 9 (9) | 4 (4)
Acute Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Maternal Anemia (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) — Maternal Anemia following intrapartum bleeding.
Bladder Trauma (Surgical and medical procedures) | 1 (1) | 0 (0) — Bladder trauma during cesarean section
Neonatal Bowel Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neonatal Cardiac Abnormalities (Congenital, familial and genetic disorders) | 2 (2) | 0 (0) — Neonatal Congenital Cardiac abnormalities such as Ventricular Septal Defect (VSD), Atrial Septal Defect (ASD) ,Patent Ductus Arteriosis (PDA)
Maternal Cellulitis (Infections and infestations) | 2 (2) | 0 (0) — maternal cellulitis at intramuscular injection site
Maternal Chorioamnionities necessitating preterm delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Neonatal Chronic Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Neonatal Congenital Hypospadium (Congenital, familial and genetic disorders) | 2 (2) | 0 (0)
Congenital Abnormality (Congenital, familial and genetic disorders) | 3 (3) | 6 (6) — neonatal congenital abnormality such as club foot, cleft palate, gastroschisis, tracheal stenosis, Hydrocele, duodenal atresia, sigmoid stricture, PDA requiring ligation.
Neonatal Cranial Synostosis (Nervous system disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (DVT) (Vascular disorders) | 1 (1) | 0 (0)
Endometritis (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Neonatal Gastroschisis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neonatal Intraventricular Hemorrhage (Stage III or IV) (Vascular disorders) | 4 (4) | 0 (0)
Maternal HELLP Syndrome (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Neonatal Hypoplastic Lung (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Intrauterine Fetal Demise (IUFD) (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0)
Neonatal Necrotizing Enterocolitis (NEC) (Gastrointestinal disorders) | 2 (2) | 3 (3)
Non-Occulusive Thrombus (Vascular disorders) | 1 (1) | 0 (0)
Peripartum Cardiomyopathy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Neonatal Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Neonatal Pneumothorax (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Neonatal Post Hemorrhagic Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Neonatal Peripheral Pulmonary Stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Severe Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Prolonged Hospitalization - Maternal Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Maternal Pyelonephritis (Renal and urinary disorders) | 2 (2) | 0 (0)
Maternal Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Compatible symptoms with diagnostic radiograph findings and positive results on blood cultures,persistent leukopenia
Neonatal Readmissions to the hospital (General disorders) | 5 (5) | 0 (0) — Neonatal readmission to the hospital after discharge = such as temperature instability, sepsis, nutritional support and apnea
Neonatal Sepsis (Infections and infestations) | 3 (3) | 5 (5) — diagnosed by clinical or laboratory findings
Maternal Supraventricular Tachycardia (SVT) (Cardiac disorders) | 1 (1) | 1 (1)
Maternal Hematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Maternal Wound Eviceration post Cesarean Section (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nectrotizing Enterocolitis (NEC) (General disorders) | 2 (2) | 3 (3)
Neonatal Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Inguinal Hernia requiring surgical repair (Surgical and medical procedures) | 0 (0) | 2 (2)
Uterine Atony (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Maternal Pyelonephritis (Renal and urinary disorders) | 2 (2) | 0 (0)
Retained Products of Conception (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Group (170HP) (N=216) | Control (Castor Oil) (N=105)
Gestational Diabetes (Metabolism and nutrition disorders) | 11 (11) | 5 (5)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 29 (29) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes